CLINICAL TRIAL: NCT01201018
Title: A Single Center, Open Label Study for Evaluation of the Safety and Efficacy of Oshadi D and Oshadi R for Cancer Treatment - A Phase I Study
Brief Title: Evaluation of the Safety and Efficacy of Oshadi D and Oshadi R for Cancer Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-DRS-P1-01
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Tumor; Cancer; Metastasis
Keywords: Tumor; cancer; metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi DR (Experimental)
  Interventions: Drug: Oshadi D, Oshadi R

INTERVENTIONS:
Drug: Oshadi D, Oshadi R — Oral administration

SUMMARY:
The study will be non randomized, open label, dose rising study in cancer patients. Cancer treatment is consisting of 2 different drugs: Oshadi D and Oshadi R that will be administered orally.

The study will include two sessions:

* A single dose period to evaluate acute toxicity of each drug
* Consecutive multiple increment dose escalation period of both drugs to determine the long-term safety, and the anticancer activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/ cytological proven solid tumor that is metastatic.
* Age > 21 years old.
* ECOG Performance status < 2.
* Documented progressive metastatic disease according to RECIST criteria.
* At least one lesion not within prior radiation field that is measurable per RECIST.
* Primary tumor must have been resected.
* Four weeks must elapse from prior therapy.
* Patient has recovered to CTCAE < Grade 1 from toxicities related to previous treatment (except non-clinically significant AEs).
* Patient must have adequate organ function.
* Sexually active fertile patients and their partners must agree to use medically accepted methods of contraception during therapy and 3 months after the last dose of the study drugs.
* Female patients of childbearing potential must have a negative pregnancy test at screening.
* Patient must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.
* Life expectancy > 6 months.

Exclusion Criteria:

* Uncontrolled Intercurrent illness or any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Current or history of hematologic malignancies.
* Patient with positive HIV serology at screening.
* Female patient who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Radiation therapy < 4 weeks prior to screening.
* Patient has received any other type of investigational agent < 4 weeks prior to screening.
* Metastatic brain or meningeal disease.
* Patient has prothrombin time/International Normalization Ration (PT/INR) or partial thromboplastin time (PTT) test results > 1.3 UNL.
* Significant swallowing disorders.
* Small bowel surgery.
* Pelvic or abdominal radiation.
* Pre-existing mal absorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption.
* Evidence of concurrent (< 5 years) second malignancy other than basal cell carcinoma of the skin or cervical carcinoma in situ.
* Mental disorders.
* Inability to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, serious adverse events occurrence | 6 months

SECONDARY OUTCOMES:
Modified "Response Evaluation Criteria in Solid Tumors" (RECIST, Appendix 3) will be used. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Avishai Sella, Prof., Principal Investigator — Assaf-Harofeh MC
Locations (1):
- Assaf-Harofeh Medical Center, Zrifin Beer-Yaakov, Israel